CLINICAL TRIAL: NCT06515912
Title: The Ketogenic Diet, Blood Lipids, and Heart Health in Healthy Adults With Differing BMI
Brief Title: Ketogenic Diet in Healthy Adults With Differing BMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KTO
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
Keywords: Ketogenic Diet
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low BMI (Experimental): BMI 18.5 - 22 kg/m^2 Intervention: Ketogenic diet 28 days
  Interventions: Other: Ketogenic Diet
- High BMI (Active Comparator): BMI 30-35 kg/m^2 Intervention: Ketogenic diet 28 days
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — A ketogenic diet with 5% carbohydrate, 18% protein, and 77% fat by percent kcal.

SUMMARY:
The goal of this clinical trial is to examine the effect of the ketogenic diet over four weeks on blood lipid levels and risk factors for heart disease in adults with a healthy BMI compared to adults with a body mass index (BMI) in the range for obesity. The main questions it aims to answer are:

* Does the ketogenic diet cause larger increases in "bad cholesterol" (low density lipoprotein-cholesterol) in adults with a healthy BMI compared to adults with BMI in the range for obesity?
* Does the ketogenic diet cause larger decreases in vascular health in adults with a healthy BMI compared to adults with BMI in the range for obesity?

Participants will:

* Consume all of the study food provided and avoid intake of non-study foods during the 28-day diet period
* Visit the metabolic kitchen daily (Monday-Friday) to pick up meals
* Attend 5 fasting visits at the Clinical Research Center for testing

DETAILED DESCRIPTION:
This is a controlled feeding study investigating if four weeks on the ketogenic diet will cause differential alterations in blood lipids and lipoproteins, vascular health as measured by fasting flow mediated dilation (FMD), and mechanistic markers of lipid metabolism in adults with normal weight when compared to adults with obesity. Outcomes will be measured at both the beginning and end of the study on two consecutive days, for a total of four clinic appointments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-45 years
2. Fasting direct LDL-C ≤100 mg/dL
3. BMI of 18.5-22 kg/m2 or 30-35 kg/m2
4. Blood pressure <140/90 mmHg
5. Fasting blood glucose <126 mg/dL
6. Fasting triglycerides <350 mg/dL
7. ≤10% change in body weight for 6 months prior to enrollment

Exclusion Criteria:

1. Have type 1 or type 2 diabetes or fasting blood glucose ≥126 mg/dL
2. Prescription of anti-hypertensive, lipid-lowering or glucose-lowering drugs
3. Intake of supplements that affect the outcomes of interest and unwilling to cease during the study period
4. Diagnosed liver, kidney, or autoimmune disease
5. Prior cardiovascular event (e.g., stroke, heart attack)
6. Current pregnancy or intention of pregnancy within the next 2 months
7. Lactation within prior 6 months
8. Follows a vegetarian or vegan diet
9. Food allergies/intolerance/sensitives/dislikes of foods included in the study menu
10. Antibiotic use within the prior 1 month
11. Oral steroid use within the prior 1 month
12. Use of tobacco or nicotine containing products within the past 6 months
13. Cancer at any site within the past 10 years (eligible if ≥10 years without recurrence) or non-melanoma skin cancer with in the past 5 years (eligible if ≥5 years without recurrence)
14. Participation in another clinical trial within 30 days of baseline
15. Currently following a restricted or weight loss diet
16. Previously consumed the ketogenic diet for more than 1 week
17. Prior bariatric surgery
18. Intake of >14 alcoholic drinks/week and/or lack of willingness to consume no alcohol while enrolled in the study and/or not willing to avoid alcohol consumption for 48 hours prior to test visits
19. Current or past eating disorder
20. Principal Investigator discretion related to the potential participant's ability to adhere to the study requirements including being able to come to the metabolic kitchen to pick-up food five days per week
21. Planning to relocate out of the State College area in the next 2 months
22. Unwilling to refrain from plasma/blood donations during the study
23. Previously diagnosed familial hypercholesterolemia
24. If a potential participant takes thyroid medicine, abnormal thyroid stimulating hormone (TSH) concentration (TSH outside of normal range of 0.5 - 4.5 mIU/L)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol concentration change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL. LDL-cholesterol will be measured directly via enzymatic assay. Change in LDL-cholesterol will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).

SECONDARY OUTCOMES:
Endothelial function - Flow Mediated Dilation (FMD) change from baseline | 4 weeks
  Assessed by fasting brachial arterial ultrasound after transient ischemia expressed in percentage (%). Change in FMD will be calculated as the end of diet measure minus the baseline measure.
Triglycerides concentration change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in triglycerides will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Total cholesterol concentration change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in total cholesterol will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
HDL-cholesterol concentration change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in HDL-cholesterol will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Concentration of LDL and triglyceride-rich lipoprotein subparticles change from baseline | 4 weeks
  Measured via Nuclear Magnetic Resonance and expressed in nmol/L. Change in concentration will be calculated as the end of diet measure minus the baseline measure.
Concentration of HDL subparticles change from baseline | 4 weeks
  Measured via Nuclear Magnetic Resonance and expressed in µmol/L. Change in concentration will be calculated as the end of diet measure minus the baseline measure.
Size of LDL, HDL, and triglyceride-rich lipoprotein particles change from baseline | 4 weeks
  Measured via Nuclear Magnetic Resonance and expressed in nm. Change in size will be calculated as the end of diet measure minus the baseline measure.
Central systolic and diastolic blood pressure change from baseline | 4 weeks
  Assessed using a SphymoCor Xcel (Atcor Medical) and expressed in mmHg. Change in blood pressures will be calculated as the end of diet measure minus the baseline measure.
Brachial systolic and diastolic blood pressure change from baseline | 4 weeks
  Assessed using a SphymoCor Xcel (Atcor Medical) and expressed in mmHg. Change in blood pressures will be calculated as the end of diet measure minus the baseline measure.
Carotid-femoral pulse wave velocity change from baseline | 4 weeks
  A measure of arterial stiffness - assessed using a SphymoCor Xcel (Atcor Medical) and expressed in meters/second. Change in pulse wave velocity will be calculated as the end of diet measure minus the baseline measure.
Serum Insulin concentration change from baseline | 4 weeks
  Assessed in a fasting blood draw and expressed in micro IU/mL. Change in insulin will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Plasma glucose concentration change from baseline | 4 weeks
  Assessed in a fasting blood draw and expressed in mg/dL. Change in glucose will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Homeostatic model assessment for insulin resistance (HOMA-IR) change from baseline | 4 weeks
  Calculated from insulin and glucose measured from a fasting blood sample. Calculated as (insulin × glucose) / 22.5. Change in HOMA-IR will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Cholesteryl ester transfer protein (CETP) activity change from baseline | 4 weeks
  Assessed in fasting plasma samples using an enzymatic activity kit. Change in CETP activity will be calculated as the end of diet measure minus the baseline measure.
Lipoprotein lipase (LPL) activity change from baseline | 4 weeks
  Assessed in fasting plasma samples using an enzymatic activity kit. Change in LPL activity will be calculated as the end of diet measure minus the baseline measure.
Angiopoietin-Like Protein 3 (ANGPTL3) concentration change from baseline | 4 weeks
  Assessed in fasting plasma samples using an ELISA kit and expressed in ng/mL. Change in ANGPTL3 concentration will be calculated as the end of diet measure minus the baseline measure.
Angiopoietin-Like Protein 4 (ANGPTL4) concentration change from baseline | 4 weeks
  Assessed in fasting plasma samples using an ELISA kit and expressed in ng/mL. Change in ANGPTL4 concentration will be calculated as the end of diet measure minus the baseline measure.
Angiopoietin-Like Protein 8 (ANGPTL8) concentration change from baseline | 4 weeks
  Assessed in fasting plasma samples using an ELISA kit and expressed in pg/mL. Change in ANGPTL8 concentration will be calculated as the end of diet measure minus the baseline measure.
Glucagon concentration change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in pg/mL. Change in glucagon concentration will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Total adiposity change from baseline | 4 weeks
  Assessed from Dual-energy X-ray absorptiometry as % body mass. Change in total adiposity will be calculated as the end of diet measure minus the baseline measure.
Estimated visceral adipose tissue change from baseline | 4 weeks
  Assessed from Dual-energy X-ray absorptiometry and calculated by software in grams (g). Change in estimated visceral adipose tissue will be calculated as the end of diet measure minus the baseline measure.
Alanine transaminase (ALT) change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in U/L. Change in ALT concentration will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Aspartate transaminase (AST) change from baseline | 4 weeks
  Assessed from fasting blood draw expressed in U/L. Change in AST concentration will be calculated as the mean of the end of diet measures (i.e., mean of day 29 and day 30 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).

OTHER OUTCOMES:
Composition of the gut microbiota | Baseline, 4 weeks
  Measured using 16 s rRNA gene sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be deposited into an open access repository once results from all pre-specified primary and secondary outcomes are published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of all pre-specified primary and secondary outcomes

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT06515912/SAP_000.pdf